CLINICAL TRIAL: NCT01037751
Title: M. D. Anderson Symptom Inventory - Ovarian Cancer: Development and Validation in Patients With Ovarian Cancer
Brief Title: M. D. Anderson Symptom Inventory - Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2009-0506
Record Dates: First submitted 2009-12-17; First posted 2009-12-23 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Ovarian Cancer
Keywords: Cancer; Symptom burden; M. D. Anderson Symptom Inventory; MDASI-Ovarian Cancer; Symptoms; Daily functioning; Symptom severity; Questionnaire; Interview
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interview + Questionnaires: 1-on-1 interview + Questionnaires, Part 1 of Study
  Interventions: Behavioral: Interview; Behavioral: Survey
- Questionnaires: Questionnaires Only, Part 2 of Study
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Interview — 1-on-1 interview with study doctor or staff member, during regularly scheduled, standard of care clinic visit taking 30 minutes.
  Groups: Interview + Questionnaires
Behavioral: Survey — Complete 3 Questionnaires during clinic visit, about 10 minutes to complete all.
  Other Names: Questionnaire

SUMMARY:
Objectives:

The objective of this study is to delineate and measure the symptom burden experienced by patients with ovarian cancer.

The Primary Aim is to develop and validate an ovarian-cancer module of the M. D. Anderson Symptom Inventory (MDASI-Ovarian Cancer) to measure the severity of multiple symptoms and the impact of these symptoms on daily functioning in patients with ovarian cancers.

The Secondary Aims are:

To develop a detailed description of symptom severity and interference with daily activities experienced by patients with ovarian cancer; To assess the impact of symptom severity on standard functioning and quality of life (QOL) measures, including Eastern Cooperative Oncology Group Performance Status (ECOG PS), Functional Assessment of Cancer Therapy-Ovary (FACT-O), and a single-item QOL scale, in patients with ovarian cancer; To define the qualitative symptom burden of patients with ovarian cancer receiving various treatments.

DETAILED DESCRIPTION:
PART 1:

Interview:

If you agree to take part in this study, you will be interviewed about what it is like to have ovarian cancer and any symptoms that you may have experienced. This will be a 1-on-1 interview with the study doctor or a member of the study staff. It will take place during 1 of your regularly scheduled, standard of care clinic visit and should take about 30 minutes to complete.

The interview will be digitally recorded. The electronic recording of the interview will be given a code number and stored on a password-protected computer at M. D. Anderson. No identifying information will be directly linked to your interview recording. Only the researcher in charge of the computer will have access to the code numbers and be able to link the interview recording to you.

Questionnaires:

After the interview, you will also complete a symptom questionnaire, a quality-of-life questionnaire, and a demographic questionnaire that asks questions about your age, race, and marital status. You will complete the questionnaires after the interview during the same clinic visit. It should take about 10 minutes to complete all 3 questionnaires.

You should contact the study doctor or study nurse right away if at any time you are experiencing severe, troublesome, or intolerable symptoms. You should also remember to rate them on the symptom questionnaire.

The questionnaires will also be given a code number and stored in a locked file cabinet at MD Anderson. No identifying information will be directly linked to your questionnaires. Only the researcher in charge of the study will have access to the code numbers and be able to link the questionnaires to you.

Length of Study:

After you have completed the interview and the questionnaires, your participation on this study will be over.

Additional Information:

Any information about your symptoms that is collected as part of this study is for research purposes only. All study materials, including the interview recording and questionnaires, will only be used for the purposes of this study and will be destroyed after the study results have been reported.

If you rate a symptom as severe on the symptom questionnaire, a study staff member will ask you if you have already told, or plan to tell your regular care doctor or nurse about the symptom. If you have not already told you regular care doctor or nurse, a study staff member will tell your regular care doctor or nurse about the symptom for you.

This is an investigational study.

Up to 15 participants will take part in this study. All will be enrolled at MD Anderson.

PART 2:

Questionnaires:

If you agree to take part in this study, you will complete the following:

1. A symptom questionnaire, 2 quality-of-life questionnaires, and a demographic questionnaire that asks questions about your age, race, and marital status. It should take about 20 minutes to complete all 4 questionnaires.
2. About 1 to 5 days after you complete the first set of questionnaires, you will be asked to complete a questionnaire either through phone interview with the study staff or through a mail-in survey . If you complete the questionnaire by mail-in survey, the study staff will give you a copy of the questionnaire and a stamped pre-addressed envelope. The questionnaire will take 5-10 minutes to complete.

You should contact the study doctor or study nurse right away if at any time you are experiencing severe, troublesome, or intolerable symptoms. You should also remember to rate them on the symptom questionnaire.

The questionnaires will be given a code number and stored in a locked file cabinet at M. D. Anderson. No identifying information will be directly linked to your questionnaires. Only the researcher in charge of the study will have access to the code numbers and be able to link the questionnaires to you.

Opinion Questionnaire:

If you are one of the first 20 patients enrolled in the study, you will be asked questions about your opinion of the symptom questionnaire. For example, you will be asked if the symptom questionnaire was easy to understand and complete, and if there were any other questions that should be included. The study staff will use your opinion to decide if changes should be made to the questionnaire or if important symptom questions are missing from the questionnaire. This questionnaire should take about 5 minutes to complete.

Length of Study:

After you have completed the questionnaires, your participation on this study will be over.

Additional Information :

Any information about your symptoms that is collected as part of this study is for research purposes only. The questionnaires will only be used for the purposes of this study and will be destroyed after the study results have been reported.

If you rate a symptom as severe on the symptom questionnaire, a study staff member will ask you if you have already told, or plan to tell your regular care doctor or nurse about the symptom. If you have not already told you regular care doctor or nurse, a study staff member will tell your regular care doctor or nurse about the symptom for you.

This is an investigational study.

Up to 128 participants will take part in this study. All will be enrolled at MD Anderson and Lyndon B. Johnson General Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients 18 years of age or older.
2. Able to speak and read English.
3. Having a diagnosis of high grade invasive epithelial ovarian cancer, peritoneal cancer or fallopian tube cancer confirmed by pathological analysis.
4. Being followed at M D Anderson Cancer Center and Lyndon B. Johnson General Hospital (LBJ Hospital).
5. Has consented to participate.
6. Has not received any current cancer treatment or prior chemotherapy in the last 30 days (phase 2 subset of 40 patients only)

Exclusion Criteria:

1) Having a medical condition or impaired performance status that would preclude participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UT MD Anderson Cancer Center ovarian cancer patients, females over the age of 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2009-12-30 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Validate ovarian-cancer module of MDASI-Ovarian Cancer to measure severity of multiple symptoms + impact of these symptoms on daily functioning in patients with ovarian cancers. | Baseline to 2 years (Patient participation done after completing Interview and Surveys during single clinic visit)

SECONDARY OUTCOMES:
Patient Rated Symptom Severity and Interference with Function (Survey Response) | Baseline to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Diane C. Bodurka, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org